CLINICAL TRIAL: NCT01234168
Title: An International, Cross Sectional, Non-interventional, Study to Assess Neuroendocrine Tumour (NET) Patients Currently Treated by Somatuline Autogel for History of Carcinoid Syndrome Associated With Episodes of Diarrhea
Brief Title: A Study to Assess Neuroendocrine Tumour (NET) Patients Currently Treated by Somatuline Autogel for History of Carcinoid Syndrome Associated With Episodes of Diarrhea
Acronym: SYMNET
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: 8-79-52030-736
Record Dates: First submitted 2010-10-20; First posted 2010-11-04 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Neuroendocrine Tumors; Carcinoid Syndrome
MeSH Terms: conditions — Neuroendocrine Tumors; Serotonin Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the protocol is to to assess subject's overall satisfaction regarding control of diarrhea. The study aims to supplement results obtained through clinical trials with data obtained from a population of patients receiving treatment with Somatuline Autogel in routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients 18 years of age and older, who have agreed to participate in the study
* Diagnosed with a Neuroendocrine tumour (NET) and receiving treatment with Somatuline Autogel

Exclusion Criteria:

* Subjects for whom there are reasons that may hinder the conduct of the study (patients who have difficulty expressing themselves or who are unable to complete the questionnaires, or with insufficient data in the their files will not be enrolled in the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out-patients
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Subject's overall satisfaction regarding control of diarrhea | Day of survey
  Use of questionnaires to assess patient satisfaction (Likert scale).

SECONDARY OUTCOMES:
Impact on daily activities of the clinical manifestations of diarrhea | Day of survey
  Use of questionnaires to assess symptom severity and impact on patient's daily activities (CGI-S).

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (57):
- Czechia (6):
  - Teaching Hospital Brno Bohunice, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - Hospital Pardubice, Pardubice
  - Teaching Hospital, Pilsen
  - Charles University, Prague
  - Teaching Hospital Na Bulovce, Prague
- France (14):
  - CHU Angers, Angers
  - Hôpital Avicenne, Bobigny
  - Hôpital Saint André, Bordeaux
  - CHU Trousseau, Chambray-lès-Tours
  - Hôpital Beaujon, Clichy
  - CHU Michallon, Grenoble
  - Hôpital Edouard Herriot, Lyon
  - CHU Timone, Marseille
  - Hôpital Archet 2, Nice
  - Hôpital du Haut Leveque, Pessac
  - Hôpital Robert Debré, Reims
  - CHU St Etienne, Saint-Priest
  - Hôpital Rangueil, Toulouse
  - Institut Gustave-Roussy, Villejuif
- Hungary (2):
  - Semmelweis University, Budapest
  - Karádi-Nagy Bt., Pécs
- Hadasit Medical Research, Jerusalem, Israel
- Italy (10):
  - Ospedale Regina Apostolorum, Albano Laziale
  - Ospedale Pesenti Fenaroli, Alzano Lombardo
  - Ospedale Civile, Castelfranco Veneto
  - Università degli Studi di Chieti, Chieti
  - Istituti Ospedalieri di Cremona, Cremona
  - Azienda Ospedaliera-Universitaria Policlinico, Modena
  - U.O.C. Malattie dell'Apparato Digerente e del Fegato, Roma
  - Unità di Endocrinologia Istituti Fisioterapici Ospitalieri, Roma
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Istituto Oncologico del Mediterraneo, Viagrande
- Poland (10):
  - Szpital Uniwersytecki im. A. Jurasza, Bydgoszcz
  - Slaskiego Uniwersytetu Medycznego, Katowice
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Szpital Uniwersytecki w Lodzi, Lodz
  - Prywatna Praktyka Lekarska, Olsztyn
  - Specjalistyczny Gabinet Lekarski, Poznan
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Szczecin
  - Niepubliczny Zaklad Opieki Zdrowotnej, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
- Spain (8):
  - Hospital Clinico Universitario de Santiago, A Coruña
  - Hospital De Cruces, Barakaldo
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital General Reina Sofia, Córdoba
  - Hospital Clinico San Carlos, Madrid
  - Hospital Xeral Cies de Vigo, Pontevedra
  - Hospital Virgen Macarena, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (6):
  - University Hospital of Wales, Cardiff
  - University Hospital, Coventry
  - University Hospital Aintree, Liverpool
  - Royal Free Hospital, London
  - Chrisite Hospital Institute, Manchester
  - Freeman Hospital, Newcastle upon Tyne

REFERENCES:
- [Derived] Ruszniewski P, Valle JW, Lombard-Bohas C, Cuthbertson DJ, Perros P, Holubec L, Delle Fave G, Smith D, Niccoli P, Maisonobe P, Atlan P, Caplin ME; SYMNET study group. Patient-reported outcomes with lanreotide Autogel/Depot for carcinoid syndrome: An international observational study. Dig Liver Dis. 2016 May;48(5):552-558. doi: 10.1016/j.dld.2015.12.013. Epub 2016 Jan 15. PMID 26917486